CLINICAL TRIAL: NCT01292746
Title: An Evaluation of the Effect of the Erchonia ML Scanner (MLS) on the Treatment of Androgenic Alopecia in Females
Brief Title: Study of the Effect of Low Level Laser Light on Hair Growth on the Female Human Scalp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and subject study compliance was difficult
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_FA001
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Female Pattern Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia ML Scanner (MLS) (Experimental): Erchonia MLS employs four diodes emitting 10 milliwatts (mW) 635 nanometer (nm) red laser light
  Interventions: Device: Erchonia MLS

INTERVENTIONS:
Device: Erchonia MLS — The Erchonia MLS administers 4 diodes of 10 milliwatts (mW) 635 nanometers (nm) red light to the scalp area for 18 minutes, 2 times each week for 12 consecutive weeks for a total of 24 treatments.

SUMMARY:
The purpose of this clinical study is to determine if the Erchonia® ML Scanner (MLS) low level laser light device can help to regrow hair on the scalp of females experiencing hair loss or thinning.

DETAILED DESCRIPTION:
Over 20 million women in the United States suffer from hair loss, and about 40% of those women are under forty years of age. The emotional aspects of hair loss for females include anxiety and depression, frustration and poor self-esteem. Androgenetic alopecia is a common cause of female balding and the most likely reason for excessive hair loss.

It is believed that light therapy of the scalp will provide an effective means to reduce hair loss and/or stimulate hair growth in females with androgenetic alopecia. Results of previous studies on low level laser therapy (LLLT) have demonstrated a variety of in vitro and in vivo effects including increased blood flow, accelerated wound healing, enhanced production of cytokines and other cellular mediators, increased cellular proliferation, among a panoply of other effects. Enhanced hair growth has been observed adjacent to treated areas in various animal models investigating the effects of LLLT. Uncontrolled studies in humans and spa-based therapies in Europe appear to show that the periodic application of low intensity light therapy reduces hair loss and appears to increase hair growth. The majority of these applications utilize light in the red and near-infrared portions of the spectrum.

The Erchonia MLS low level laser is being evaluated for its potential to improve the quality and quantity of hair on the female scalp. This may improve the quality of life as a result of improved self-image and may potentially delay or reduce the need for surgical procedures such as hair transplantation. A successful local therapy would mitigate or reduce the need for systemic agents such as minoxidil and finasteride, thereby minimizing the potential side effects of these therapies.

ELIGIBILITY:
Inclusion Criteria:

* Female pattern androgenic alopecia defined as:

  * discernable decrease in hair density on the top of the scalp relative to the sides and back of the scalp (ii) classifications I-3, I-4, II-1, II-2 according to the Ludwig and Savin Hair Loss Scale
* Notable hair loss/thinning onset within the past five years.
* Progressive/active hair loss/thinning within the last 12 months.
* Skin type I through IV according to the Fitzpatrick Skin Type Scale.
* Healthy, balanced scalp, determined as one that shows no indication of notable: dryness, flaking, dandruff (pityriasis), redness, irritation, inflammation, itching, greasy/oily texture, odor, lesions, scalp acne or other significant dermatological conditions.
* PI or P2 on the American Society of Anesthesiologists (ASA) Physical Status Classification System.
* Willing and able to maintain same hair style, length, color and hair care regimen throughout study participation.

Exclusion Criteria:

* Hair loss attributable to one or more of the following conditions: tinea capsitis, secondary syphilis, discoid lupus erythematosus: Inflammation, alopecia areata, trichotillomania, telogen effluvium, anagen effluvium, traumatic alopecia.
* Use of any of the following medications presently or during the prior 6 months: minoxidil, finasteride (or any other 5ᾳ-reductase inhibitor medications),medication with anti-androgenic properties (e.g. cyproterone, spironolactone, ketoconazole, flutamide and bicalutamide),topical estrogens, progesterone, tamoxifen, anabolic steroids, medications that can potentially cause hypertrichosis (e.g. ciclosporin, diazoxide, phenytoin and psoralens), oral glucocorticoids (inhaled glucocorticoids permitted), lithium, phenothiazines.
* Current use of other prescription and/or over-the-counter products known to affect hair growth and distribution (e.g. saw palmetto, fish oil, corticosteroids, antineoplastic agents, beta blockers, diazoxide, heparin, verapamil, warfarin, etc.).
* Medical, physical, or other contraindications for, or sensitivity to, light therapy (e.g. porphyria, photosensitizing drug therapies).
* Taking Hormonal Replacement Therapy.
* Conditions that may worsen with light therapy.
* History of poor wound healing.
* History of keloid formation.
* Prior hair restoration/transplantation surgery.
* Prior scalp reduction procedure(s).
* Other surgery to the scalp region (e.g. to remove a skin cancer lesion).
* Active skin infection, wound, or other external trauma to the scalp evaluation area.
* Active malignancy or any malignancy in the past five years in the scalp evaluation area.
* Dermatological condition (dermatitis, eczema, psoriasis, etc.) of the scalp other than female pattern hair loss.
* Significant scarring (e.g. from burns) in the scalp evaluation area.
* History of thyroid condition that may influence hair growth and loss.
* Underlying medical condition(s) known to adversely affect hair growth or hair pattern, such as HIV, connective tissue disease, inflammatory bowel disease.
* Current hair weaves.
* Use of non-breathable wigs.
* Hairstyle is a "buzz" cut, defined as hair cut to less than one inch in length.
* Tattooing of the scalp target evaluation area.
* Subject is pregnant, nursing, planning a pregnancy, or less than six months postpartum.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to record study measurements.
* Involvement in litigation/receiving disability benefits related in any way to the parameters of the study.
* Participation in research in the past 30 days.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Thaxton, MD, FACOG, Principal Investigator
Locations (1):
- Advanced Gynecology Specialists of Georgia, Evans, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia MLS: Erchonia MLS employs four diodes emitting 10 milliwatts (mW) 635 nanometer (nm) red laser light.
Period: Overall Study
Arm/Group | Erchonia MLS
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia MLS
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Non-Vellus Terminal Hair Count [Mean (Standard Deviation); unit: hairs/cm2] — Non-vellus terminal hair count per centimeter squared (cm2) was calculated by independent evaluator analysis employing digital photograph images and macroimage analysis software
  hairs/cm2 | 171.57 (60.78)

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-vellus Terminal Hair Count Across a 3 cm Diameter Scalp Area
Description: Non-vellus terminal hair count was calculated across a tattooed 3 cm diameter scalp area from digital photographs of the area by independent blinded evaluator employing macroimage analysis software.
Time Frame: Baseline and 13 Weeks
Measure: Mean (Standard Deviation); unit: hairs/cm2
Arm/Group | Erchonia MLS
Number analyzed (Participants) | 14
hairs/cm2 | 10.93 (13.90)
Statistical Analysis 1: Comparison: Erchonia MLS; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; 2 sided t-test for correlated samples

ADVERSE EVENTS:
Time Frame: 13 Weeks
Arm/Group | Erchonia MLS
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No